CLINICAL TRIAL: NCT01807988
Title: Regional Study of Internet-based Relapse Prevention as an Adjunct to Partially Successful Antidepressant Medication
Brief Title: Internetbased Relapse Prevention for Partially Remitted Depression
Acronym: ISAK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Örebro County Council (Other Government)
Collaborators: Uppsala University (Other); Uppsala County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Fredrik Holländare, Clinical Psychologist, PhD, Örebro County Council
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012/488
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Depression
Keywords: Relapse, Recurrence, Depression, Internet, Sick-leave
MeSH Terms: conditions — Depression; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- iCBT (Experimental): Internetbased cognitive behavior therapy (iCBT) aimed att preventing relapse into major depression.
  Interventions: Behavioral: iCBT
- Control group (No Intervention): The control group in the study will fill out questionnaires every month and will be interviewed every month to detect any relapses. They will also receive feedback on there self-reported symptoms.

INTERVENTIONS:
Behavioral: iCBT — Internetbased cognitive behavior therapy (iCBT) contains interventions that will help the participant to change her behavior to experience more positive reinforcement in daily life and also to challenge her negative patterns of thought. There are also information and exercices to improve sleep, increase physical activity, train mindfulness, handle anxiety and to learn about depression.
  Arms: iCBT

SUMMARY:
The main purpose of the study is to test whether Internet-based relapse prevention plus medication has a better protective effect compared to medication only, for persons with residual depressive symptoms who are currently in paid employment or in education. We hypothesise that during the two years following the intervention:

* The persons in the group receiving Internet-based relapse prevention plus medication will be absent from work for fewer days due to sick-leave compared to those in the medication-only group.
* Fewer persons in the group receiving Internet-based relapse prevention + medication will experience long term sick-leave (60 days or more) compared to those in the medication-only group.
* The persons in the group receiving Internet-based relapse prevention plus medication will suffer fewer depressive relapses compared to those in the medication-only group.
* At follow-up, the persons in the group receiving Internet-based relapse prevention plus medication will have higher health related quality of life and lower levels of depressive symptoms compared to those in the medication-only group.

ELIGIBILITY:
Inclusion Criteria:

* Mild residual depressive symptoms (7-19 on the MADRS-S).
* A history of at least one episode of Major Depression.
* Currently in (at least) half-time employment, self-employment or education.
* Taking a stable (since one month) and therapeutic dosage of antidepressant medication
* Being able to read and write Swedish
* Having access to the internet

Exclusion Criteria:

* Fulfilling the criteria for Major depression
* Psychosis
* Substance abuse
* Suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Days absent from work due to sick leave | 24 month follow up
  The total number of days that a participant has been absent from work due to sick leave (any cause). Data will be collected from the National Insurance Agency at the end of the study.
Change in self-reported sick leave days | After 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24 months
  Self-reported number of sick leave days during the study will be collected cumulatively every month during the study time and summarised after 24 months.
Change in diagnostic status | After 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24 months
  Change in diagnostic status (depressive relapse) will be assessed in a telephone interview every month during the study. The definition of a relapse is to fulfill the diagnostic criteria for major depression according to the DSM-IV at any time after the study start.
Change in depressive symptoms | After 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24 months
  Change in depressive symptoms will be measured by an internetbased version of the Montgomery-Asberg Depression Rating Scale - Self rated. The patient will fill out the questionnaire every month.

SECONDARY OUTCOMES:
Change in health related quality of life | After 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24 months
  Health related quality of life will be measured by an internetbased version of the EQ-5D. The questionnaire will be filled out every month.
Change in costs associated with illness | Pre- and post treatment, after 12 and 24 months
  Change in costs will be measured by an internetbased version of the self-assessment scale Trimbos/iMTA questionnaire on Costs associated with Psychiatric illness (TIC-P).

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Psychiatric Research Centre, Örebro
  - Psychiatric Clinic in Uppsala, Uppsala